CLINICAL TRIAL: NCT00563316
Title: A Phase I, Open-label Study to Determine the Effect of Panitumumab on the Pharmacokinetics of Irinotecan in Subjects With Unresectable Metastatic Colorectal Cancer
Brief Title: Effect of Panitumumab on the Pharmacokinetics of Irinotecan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20062010
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; chemotherapy; cancer; metastatic; irinotecan; EGFr; epidermal growth factor
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Panitumumab; Irinotecan

ARMS (1):
- Panitumumab + Irinotecan (Experimental): Participants received panitumumab 6 mg/kg and irinotecan 180 mg/m² administered by intravenous (IV) infusion every 2 weeks until disease progression or intolerance of panitumumab, irinotecan or both.
  Interventions: Drug: Panitumumab; Drug: Irinotecan

INTERVENTIONS:
Drug: Panitumumab — The first infusion of panitumumab will occur on Cycle 1 Day 4. On Cycle 2 Day 1, panitumumab will be administered on the same day as irinotecan and every 2 weeks thereafter.
  Other Names: Vectibix
Drug: Irinotecan — The first infusion of irinotecan will occur on Cycle 1 Day 1. Irinotecan will be administered on the same day as panitumumab on Cycle 2 Day 1 and every 2 weeks thereafter.
  Other Names: Camptosar

SUMMARY:
The primary objective of this study is to determine if panitumumab affects the pharmacokinetic (PK) profile of irinotecan.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed unresectable metastatic colorectal cancer (mCRC) which has progressed on at least one prior 5-fluorouracil (5FU)-containing chemotherapy regimen
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy of ≥ 3 months as documented by the investigator
* Baseline actual body weight ≤ 160 kg
* Competent to comprehend, sign, and date a written Institutional Review Board (IRB) approved informed consent form before any study-specific procedures are performed

Exclusion Criteria:

* Treatment with radiotherapy ≤ 14 days before enrollment. Patients must have recovered from all radiotherapy-related toxicities
* Known presence of central nervous systems (CNS) metastases
* Any prior malignancy (except for non-melanomatous skin cancer or in situ cervical cancer) other than the study disease, unless treated with curative intent with no evidence of disease ≤ 2 years before enrollment
* History of interstitial lung disease (eg, pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest computed tomography (CT) scan
* Active inflammatory bowel disease or other bowel disease causing chronic diarrhea (defined as > Common Terminology Criteria for Adverse Events (CTCAE version 3) grade 2
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrollment
* UGT1A1*28 TA7/7, TA7/8, TA8/8 genetic polymorphisms; Gilbert's Disease
* Treatment with CYP3A4 enzyme inhibiting or inducing medications ≤ 2 weeks before enrollment
* Prior anti-epidermal growth factor receptor (EGFr) antibody therapy (eg, cetuximab) or treatment with small molecule EGFr inhibitors (eg, gefitinib, erlotinib, lapatinib)
* Systemic chemotherapy, hormonal therapy, immunotherapy, or experimental or approved proteins/antibodies (eg, bevacizumab) ≤ 30 days before enrollment
* Subjects requiring immunosuppressive agents (eg, methotrexate and cyclosporine), however corticosteroids are allowed
* Major surgery < 28 days prior to enrollment or minor surgery (excluding catheter placement) < 14 days before enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (6):
- United States (4):
  - Research Site, Billings, Montana
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
- Canada (2):
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario

REFERENCES:
- [Background] Yang BB, Wu CY, Chen E, Infante JR, Chen A, Gao B, Smith B, Litten J, Kennecke H. Pharmacokinetics of Irinotecan With and Without Panitumumab Coadministration in Patients With Metastatic Colorectal Cancer. Clin Pharmacol Drug Dev. 2013 Jul;2(3):205-12. doi: 10.1002/cpdd.35. Epub 2013 May 15. PMID 27121781
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 6 sites in the United States and Canada. The first patient enrolled on 28 March 2008 and the last patient enrolled on 30 January 2009. Results are reported up until the data cut-off date of 16 July 2009.
Period: Overall Study
Arm/Group | Panitumumab + Irinotecan
Started | 28
Received Investigational Product | 27
Completed | 16
Not Completed | 12
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 2
Not completed — Death | 1
Not completed — On-going in study as of 16 July 2009. | 5
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set (all participants who received at least 1 dose of panitumumab or irinotecan)
Arm/Group | Panitumumab + Irinotecan
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 18
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 17
  Black or African American | 0
  Hispanic or Latino | 0
  Asian | 8
  Japanese | 1
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  Aborigine | 0
  Other | 1
Primary Tumor Type [Number; unit: participants]
  Colon Cancer | 17
  Rectal Cancer | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Irinotecan
Description: To analyze the effect, if any, that panitumumab had on the pharmacokinetics of irinotecan, the Cmax of irinotecan administered alone (Cycle 1) and with concomitant panitumumab (Cycle 2) was measured. Plasma samples were assayed by a validated high performance liquid chromatography (HPLC)-fluorescence method for the measurement of irinotecan. The lower limit of quantitation (LLOQ) was 2 ng/mL.
Time Frame: Predose and at 10 minutes, and 0.5, 1, 2, 4, 8, 24, 48, and 72 hours after the end of the irinotecan infusion at cycle 1 (irinotecan alone, week 1 day 1) and cycle 2 (irinotecan with panitumumab, week 3, day 1).
Population: The pharmacokinetic analysis set included all participants who received panitumumab 6 mg/kg and irinotecan 180 mg/m² without dose reductions or delays and who completed the blood sample collection for pharmacokinetic analysis during cycles 1 and 2.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panitumumab + Irinotecan
Number analyzed (Participants) | 19
ng/mL
  Cycle 1 | 1570 (321)
  Cycle 2 | 1570 (520)
Statistical Analysis 1: Comparison: Panitumumab + Irinotecan; Test type: Non-Inferiority or Equivalence — It would be concluded that panitumumab did not have a clinically important effect on the pharmacokinetics of irinotecan if the 90% confidence intervals of the ratio of geometric means for the Cmax and AUC values for irinotecan with and without concomitant panitumumab administration fell within the interval of 70% to 143%; Least Squares Geometric Mean Ratio = 0.980, 90% CI 2-sided [0.894 to 1.074] — Ratio of Cycle 2 : Cycle 1

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From the Time of Dosing to Infinity (AUCinf) for Irinotecan
Description: To analyze the effect, if any, that panitumumab had on the pharmacokinetics of irinotecan, the AUCinf of irinotecan administered alone (Cycle 1) and with concomitant panitumumab (Cycle 2) was measured.
Time Frame: as for outcome 1
Population: The pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Panitumumab + Irinotecan
Number analyzed (Participants) | 19
hr*ng/mL
  Cycle 1 | 12000 (4350)
  Cycle 2 | 10700 (3930)
Statistical Analysis 1: Comparison: Panitumumab + Irinotecan; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Least Squares Geometric Mean Ratio = 0.898, 90% CI 2-sided [0.819 to 0.985] — Ratio of Cycle 2 : Cycle 1

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From the Time of the Last Quantifiable Concentration (AUClast) for Irinotecan
Description: To analyze the effect, if any, that panitumumab had on the pharmacokinetics of irinotecan, the AUClast of irinotecan administered alone (Cycle 1) and with concomitant panitumumab (Cycle 2) was measured.
Time Frame: as for outcome 1
Population: The pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Panitumumab + Irinotecan
Number analyzed (Participants) | 19
hr*ng/mL
  Cycle 1 | 11900 (4290)
  Cycle 2 | 10600 (3870)
Statistical Analysis 1: Comparison: Panitumumab + Irinotecan; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Least Squares Geometric Mean Ratio = 0.897, 90% CI 2-sided [0.818 to 0.983] — Ratio of Cycle 2 : Cycle 1

4. Primary Outcome: Number of Participants With Clinically Significant Adverse Events (AEs)
Description: Adverse events of special interest include infusion reactions, integument toxicities, diarrhea, stomatitis, hypomagnesemia, and pulmonary, vascular, and cardiac toxicities. Infusion reactions were defined as 1. Prespecified signs and symptoms indicating a possible infusion reaction (derived from Common Terminology Criteria for Adverse Events (CTCAE) definitions of allergic reaction/hypersensitivity and cytokine release syndrome/acute infusion reaction) with onset day coincident with any study drug infusion and which resolved the day of, or the day after, onset; 2. incidence of AE with terms consistent with the panitumumab US package insert (USPI) (any event within 24 hours of an infusion during the clinical study described as allergic reaction or anaphylactoid reaction, or any event occurring on the first day of dosing described as allergic reaction, anaphylactoid reaction, fever, chills, or dyspnea).
  Data are summarized overall and by treatment phase.
Time Frame: The reporting time frame for Adverse Events is from first dose date to 30 days since the last dose date, until the data cut-off date of 16 July 2009. The median time frame is 5.7 months.
Population: All treated participants
Measure: Number; unit: participants
Groups:
- Treatment Phase 1: Cycle 1 Irinotecan - After irinotecan administration, but before panitumumab administration.
- Treatment Phase 2: Cycle 1 Irinotecan and Panitumumab - After first panitumumab administration until the start of Cycle 2.
- Treatment Phase 3: Cycle 2 Irinotecan and Panitumumab - After irinotecan administration until 72 hours after administration.
- Treatment Phase 4: All Other - 72 hours after administration of irinotecan in Cycle 2 until end of study.
Arm/Group | Panitumumab + Irinotecan | Treatment Phase 1 | Treatment Phase 2 | Treatment Phase 3 | Treatment Phase 4
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
participants
  Any adverse events of Interest | 27 | 5 | 26 | 9 | 26
  Integument Toxicities | 25 | 0 | 24 | 2 | 24
  Diarrhea | 23 | 2 | 12 | 4 | 20
  Hypomagnesemia | 13 | 0 | 1 | 0 | 13
  Stomatitis/Oral Mucositis | 13 | 0 | 6 | 0 | 8
  Pulmonary Toxicity | 9 | 0 | 4 | 1 | 7
  Infusion Reaction CTCAE | 8 | 2 | 0 | 5 | 4
  Infusion Reaction USPI | 2 | 1 | 0 | 0 | 1
  Vascular Toxicity | 5 | 0 | 2 | 0 | 3
  Neuro Toxicities | 3 | 0 | 1 | 1 | 1
  Cardiac Toxicity | 2 | 1 | 0 | 0 | 2
  Hematological Toxicities | 2 | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: The reporting time frame for Adverse Events is from first dose date to 30 days since the last dose date, until the data cut-off date of 16 July 2009. The median time frame is 5.7 months.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Panitumumab With Irinotecan: Participants received panitumumab 6 mg/kg and irinotecan 180 mg/m² administered by intravenous (IV) infusion every 2 weeks until disease progression or intolerance of panitumumab, irinotecan or both.
Arm/Group | Panitumumab With Irinotecan
Serious Adverse Events (participants affected / at risk) | 4/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab With Irinotecan (N=27)
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Gait disturbance (General disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab With Irinotecan (N=27)
Anaemia (Blood and lymphatic system disorders) | 2
Blepharitis (Eye disorders) | 2
Conjunctivitis (Eye disorders) | 2
Dry eye (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain lower (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Chapped lips (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 23
Dyspepsia (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 12
Stomatitis (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 9
Chest pain (General disorders) | 2
Chills (General disorders) | 2
Fatigue (General disorders) | 25
Infusion related reaction (General disorders) | 2
Mucosal inflammation (General disorders) | 6
Non-cardiac chest pain (General disorders) | 2
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 2
Pyrexia (General disorders) | 5
Xerosis (General disorders) | 9
Paronychia (Infections and infestations) | 10
Rhinitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 2
Weight decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 9
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 13
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Cholinergic syndrome (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 8
Urinary hesitation (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 8
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 19
Dry skin (Skin and subcutaneous tissue disorders) | 7
Nail disorder (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 6
Skin fissures (Skin and subcutaneous tissue disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.